CLINICAL TRIAL: NCT02166372
Title: Taiwan Diabesity Study:Comparison With Mild Obese T2DM Patients Who Under Metabolic Surgery
Acronym: TDS
Status: Recruiting | Type: Observational
Sponsor: Min-Sheng General Hospital (Other)
Responsible Party: Principal Investigator, WEI-CHENG YAO, Professor, Min-Sheng General Hospital
Other Study IDs: MSIRB2014009
Record Dates: First submitted 2014-06-16; First posted 2014-06-18 (Estimated); Last update posted 2014-06-18 (Estimated); Status verified 2014-06

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Obese diabetic patients: Diabetic patients with BMI over 25 Age 20 to 67 Diabetes medically controlled at our center for at least six months
  Interventions: Other: Observation of natural course of Diabetes Mellitus Type 2

INTERVENTIONS:
Other: Observation of natural course of Diabetes Mellitus Type 2

SUMMARY:
T2DM has become a major health burden for our society. More and more data support the relative effectiveness of gastrointestinal metabolic surgery, known as bariatric surgery, in the remission of T2DM of BMI less35. The metabolic surgery guidelines of IDF recommend BMI over 27.5 in Asia.

The evidence reviewed above strongly points to the need for a large randomized, controlled trial to evaluate the risks and benefits of obesity surgery in the treatment of type 2 diabetes Mellitus. This study is expected to provide very significant findings about the natural course of diabetes in obese diabetic patients.

DETAILED DESCRIPTION:
This study will recruit 200 obese T2DM patients at MSGH, for a total of 1000 in Taiwan. The inclusion criteria are those with T2DM more than 6 months, under medical management in diabetes center, BMI over 25, age between 20 and 67 years. The goals of this study are to evaluate the nature course of the diabetes for 10 years. The primary outcomes for the treatment will be assessed every year after intervention and will be composite of CVD risk factor; specifically, the proportion of patients with HbA1c < 7%, LDL cholesterol < 100 mg/dl and systolic blood pressure < 140 mmHg.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic Mellitus Type 2 medically controlled at Diabetes Center for at least six months
* BMI over 25
* age between 20 and 67

Exclusion Criteria:

* Diagnosed with cancer within past five years
* HIV positive
* Active TB patients
* CV events in past six months
* serum cretinine over 2.0 mg/dl
* C-peptide bellow 1.0 ng/ml in past three months
* Diabetic retinopathy; vision bellow 0.1
* Cushing's syndrome
* History of organ transplant
* History of bariatric surgery
* History of alcohol or drug dependency in past five years
* Psychological problems likely to interfere with adherence to protocol

Ages: 20 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diabetic patients in Taiwan
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2014-03; Primary Completion 2024-12 (Estimated); Study Completion 2034-12 (Estimated)

PRIMARY OUTCOMES:
Evaluate the natural course of the diabetes of obese patients over a period of 10 years | ten years

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Jei Lee, MD PhD, Principal Investigator — Min-Sheng General Hospital; National Taiwan University Hospital
Locations (1):
- Min-Sheng General Hospital, Taoyuan, Taiwan